CLINICAL TRIAL: NCT00508287
Title: Randomized, Placebo-Controlled, Single-Dose, Crossover Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-686117 in Subjects With Type 2 Diabetes
Brief Title: Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-686117 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MB110-005
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BMS 686117; Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: BMS-686117
- B (Active Comparator)
  Interventions: Drug: Byetta
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-686117 — Injection solution, Subcutaneous, 1 mg, Once daily, Single dose.
  Arms: A
Drug: Byetta — Injection solution, Subcutaneous, 5 mcg, Once daily, Single dose.
  Arms: B
Drug: Placebo — Injection solution, Subcutaneous, 1 mg, Once daily, Single dose.
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics and pharmacodynamics of single doses of BMS-686117

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes for ≥ 3 months treated with metformin, thiazolidinedione, or sulfonylurea (either monotherapy or combination) or diet alone (drug naïve)
* Fasting plasma glucose: 126 - 240 mg/dL
* Hemoglobin A1c: 6 - 10%
* Estimated CrCl ≥ 60 mL/min
* ALT ≤ 1.5 x ULN and total bilirubin ≤ 2 x ULN
* Stable and well controlled hypertension and/or dyslipidemia
* Concomitant medications used for hypertension and/or dyslipidemia, thyroid hormone replacement therapy and low dose aspirin will be allowed if stable for at least 6 weeks

Exclusion Criteria:

* Women of childbearing potential
* Symptomatic diabetes with polyuria and/or polydipsia
* History of diabetic ketoacidosis or hyperosmolar nonketotic syndrome
* History of renal disease including diabetic nephropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of adverse events | from subject enrollment to study discharge

SECONDARY OUTCOMES:
PK parameters: Cmax, Tmax, AUC(0-24h), AUC(INF) and T-HALF | from pre-dose to 24 hrs post-dose
PD Measures: Fasting and postprandial serum glucose (AUC), serum insulin, and plasma glucagon concentrations. Acetaminophen plasma concentrations will be measured after a single dose of acetaminophen | from pre-dose to 9 hrs post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Elite Research Institute, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center For Clinical Research, Knoxville, Tennessee